CLINICAL TRIAL: NCT03679533
Title: The Impact of Cranberries on the Microbiome and the Brain in Healthy Ageing: A Feasibility Intervention
Brief Title: The Impact of Cranberries On the Microbiome and the Brain in Healthy Ageing sTudy (COMBAT)
Acronym: COMBAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of East Anglia (Other)
Collaborators: Clinical Research and Trials Unit (Norfolk & Norwich University Hospital, UK) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: R204719
Record Dates: First submitted 2018-06-15; First posted 2018-09-20 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Aging; Cognitive Decline
Keywords: Cognition; Ageing; Nutrition; Microbiome; Flavonoids
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Double-blind placebo-controlled parallel intervention
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Cranberry Study Food (Active Comparator)
  Interventions: Dietary Supplement: Freeze-Dried Cranberry Powder
- Placebo Study Food (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Freeze-Dried Cranberry Powder — Freeze-dried cranberry powder (or matched placebo), approximating 500mg active flavonoids per day, taken twice daily for 12 weeks.
  Arms: Active Cranberry Study Food
Dietary Supplement: Placebo — Placebo food powder matched for taste, colour, energy and macronutrient content to the active cranberry powder.
  Arms: Placebo Study Food

SUMMARY:
Tremendous progress has been made in characterizing the interactions between the central nervous system and the gastrointestinal tract. This concept of a gut-brain axis suggests that influencing bacteria in the gut is a promising approach for developing new ways of benefiting brain function. This is particularly relevant for an ageing population for which cognitive decline is a common symptom and can be an indicator for the development of neurodegenerative conditions such as dementia. There is good evidence already that nutrition can delay the development of cognitive decline in ageing, in particular for ageing-sensitive brain regions such as the medial temporal lobe, however this has been little explored for cranberry intake. Cranberries are high in plant-derived nutrients called polyphenols, which have been suggested to promote brain function and protect against disease-causing mechanisms. In the proposed project we will pioneer work to investigate the impact of cranberry intake on gut bacteria and how it relates to cognitive performance in ageing and associated regions in the brain.

This study is being conducted by Chief Investigators Dr David Vauzour and Prof Michael Hornberger at the University of East Anglia. Sixty participants (i.e. n=30 control and treatment groups) aged 50-80 years old, with no memory complaints will be recruited for this 12-week double-blind placebo-controlled parallel intervention of cranberry flavonoids. Freeze-dried cranberry or a matched placebo will be taken twice daily for the duration of the trial. Blood, urine and faecal samples will be collected for microbiome, DNA, biochemical and nutritional analysis. Participants will also undergo cognitive testing, as well as MRI scanning to detect changes in brain physiology.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 50 and 80 years old.
* Willing and able to provide written informed consent.
* Fluent in written and spoken English.
* Normal or corrected to normal vision and hearing.
* Understands and is willing and able to comply with all study procedures.

Exclusion Criteria:

* Diagnosis of any form of dementia or significant neurological condition.
* Significant memory complaints.
* Past history or MRI evidence of brain damage, including significant trauma, stroke, learning difficulties or serious neurological disorder, including a loss of consciousness for more than 24 hours.
* Currently smoking or ceased smoking less than 6 months ago.
* Chronic fatigue syndrome, liver disease, diabetes mellitus, or gall bladder abnormalities.
* History of alcohol or drug dependency.
* Clinically diagnosed psychiatric disorder.
* Existing diagnosed gastrointestinal disorders likely to impact on absorption of flavonoids.
* Known allergy to the intervention supplement.
* Any significant medical condition likely to affect participation.
* Currently a participant or have been a participant in any other study involving an investigational product within the last 4 weeks.
* Uncontrolled hypertension (systolic blood pressure >140mmHg, diastolic blood pressure >90mmHg).
* Major cardiovascular event, such as myocardial infarction, within the last 12 months.
* On a stable prescription of blood pressure lowering medication or non-steroidal anti-inflammatory drugs. for fewer than 2 months.
* Prescribed anti-coagulant/blood thinning medication (eg. warfarin).
* Taking flavonoid containing supplements (and unwilling to cease intake during, and 1 month preceding the trial) or unwilling to maintain existing intake of other supplements.
* High flavonoid intake defined as > 15 portions of flavonoid rich foods per day
* Are currently taking medication or supplements which have a significant impact on the outcome measures.

In addition, any participants with claustrophobia will not be invited to participate in the neuroimaging component of the study. Likewise for metal implants, e.g. pacemaker that precludes MRI.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-10-02 (Actual); Primary Completion 2020-05-22 (Actual); Study Completion 2020-05-22 (Actual)

PRIMARY OUTCOMES:
Gut microflora speciation and metabolism | 12 weeks
  Measured in faecal and serum samples.
Change in volumes of hippocampus and other key brain structures | 12 weeks
  Structural magnetic resonance imaging
Change in cerebrovascular blood flow | 12 weeks
  Measured using spectroscopy
Change in global cognition | 12 weeks
  Global cognition to be measured using the Addenbrooke's Cognitive Examination - III, from 0-100, with higher scores indicating better global cognitive performance.
Change in spatial navigation abilities | 12 weeks
  The Supermarket Test, with outcomes including accurate reporting of starting direction, and accurate indication of end position and direction.
Change in executive function and attention | 12 weeks
  Trail Making Test, with scores including time taken to complete and number of errors made.
Change in memory performance | 12 weeks
  The Rey Complex Figure Test, with outcomes including time taken to complete copy, accuracy out of a possible 36 of copy and accuracy out of 36 of 3-minute recall.
Change in spatial navigation abilities | 12 weeks
  SeaHero Quest Test, with outcomes including time taken to complete, accuracy of path taken and number of errors made.
Change in executive function and attention | 12 Weeks
  Digit Span Backwards, scored out of a possible 14 for numbers recited backwards in the correct order.
Change in presence of circulating inflammatory biomarkers (hs-CRP) | 12 weeks
  Blood samples analysed for presence of inflammatory cytokines
Change in circulating biomarkers of neuronal functioning and cognitive decline (BDNF) | 12 weeks
  Blood samples analysed for presence of circulating biomarkers of neural function
Change in circulating biomarkers of lipid metabolism (total-, HDL-, LDL-cholesterol) | 12 weeks
  Blood samples analysed for presence of circulating biomarkers of lipid metabolism
Change in circulating biomarkers of lipid metabolism (triglycerides) | 12 weeks
  Blood samples analysed for presence of circulating biomarkers of lipid metabolism

SECONDARY OUTCOMES:
Changes in energy expenditure and sleep | 12 weeks
  Actigraphs to be used to measure changes in activity and sleep patterns of participants.
Genetics related to neurodegenerative disease | Baseline
  Blood samples to be analysed for genes associated with neurodegenerative disease and dementia (eg. C9ORF72, APOE-4)
Biomarkers of gut permability and endotoxemia (LPS) | 12 weeks
  Blood serum/plasma samples to be analysed for presence of lipopolysaccharide (LPS) as a biomarker of gut permability and possible endotoxemia
Levels of sunlight exposure | Baseline, Follow-up
  Self-reported levels of daily sunlight exposure to be measured using a brief questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: David Vauzour, PhD, Principal Investigator — University of East Anglia; Michael Hornberger, PhD, Principal Investigator — University of East Anglia
Locations (1):
- University of East Anglia, Norwich, Norfolk, United Kingdom

REFERENCES:
- [Derived] Flanagan E, Cameron D, Sobhan R, Wong C, Pontifex MG, Tosi N, Mena P, Del Rio D, Sami S, Narbad A, Muller M, Hornberger M, Vauzour D. Chronic Consumption of Cranberries (Vaccinium macrocarpon) for 12 Weeks Improves Episodic Memory and Regional Brain Perfusion in Healthy Older Adults: A Randomised, Placebo-Controlled, Parallel-Groups Feasibility Study. Front Nutr. 2022 May 19;9:849902. doi: 10.3389/fnut.2022.849902. eCollection 2022. PMID 35662954